CLINICAL TRIAL: NCT00003673
Title: A Study of the Safety of CMA-676 in Treatment of Elderly Patients With Acute Myeloid Leukemia (AML) in First Relapse
Brief Title: CMA-676 in Treating Older Patients With Acute Myeloid Leukemia in First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: W-AR-0903B1-203-US; CDR0000066771; NCI-V98-1497
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Drug Therapy; Gemtuzumab

INTERVENTIONS:
Drug: chemotherapy
Drug: gemtuzumab ozogamicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of CMA-676 in treating older patients who have acute myeloid leukemia that has recurred for the first time following at least 3 months of complete remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of CMA-676 in elderly patients with acute myeloid leukemia in first relapse in terms of the number of patients attaining a complete remission. II. Assess the safety of CMA-676 in this patient population.

OUTLINE: This is an open label, single arm, multicenter study. Patients receive 1 course of CMA-676 IV over 2 hours on day 1 followed by a 6 hour observation period. Patients may receive 1 additional course of therapy 15 to 28 days later. There is a 28 day follow-up period after the last dose of study medication. Patients are followed for an additional 6 months, then every 3 months for 18 months, and then every 6 months until relapse and/or death.

PROJECTED ACCRUAL: A total of 23-55 patients will be accrued for this study within 12 months. Enrollment will then be extended for up to an additional 55 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: CD33 positive acute myeloid leukemia in first relapse At least 3 months of complete remission No history of a secondary leukemia evolving from a known prior myelodysplastic syndrome or resulting from exposure to chemotherapy or toxins No active CNS leukemia

PATIENT CHARACTERISTICS: Age: 60 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC less than 30,000/mm3 at time of CMA-676 administration Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 3.0 mg/dL Cardiovascular: No uncontrolled cardiac disease Pulmonary: No uncontrolled pulmonary disease Other: No other active malignancy No uncontrolled, life-threatening infections Able to obtain bone marrow aspirate HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow and peripheral blood stem cells transplantation No prior anti-CD33 antibody therapy Chemotherapy: Prior cytotoxic chemotherapy for AML allowed No prior chemotherapy for AML in first relapse except hydroxyurea At least 24 hours since prior hydroxyurea Recovered from prior antineoplastic therapy (except alopecia) No concurrent cytotoxic chemotherapy Endocrine therapy: No concurrent immunosuppressive therapy Radiotherapy: Not specified Surgery: Not specified Other: At least 4 weeks since prior investigational agents No other concurrent antileukemic therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 1998-03; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stanley Berger, MD, Study Chair — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (10):
- United States (10):
  - Arizona Cancer Center, Tucson, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Lang K, Menzin J, Earle CC, Mallick R. Outcomes in patients treated with gemtuzumab ozogamicin for relapsed acute myelogenous leukemia. Am J Health Syst Pharm. 2002 May 15;59(10):941-8. doi: 10.1093/ajhp/59.10.941. PMID 12040733
- [Background] Larson RA, Boogaerts M, Estey E, Karanes C, Stadtmauer EA, Sievers EL, Mineur P, Bennett JM, Berger MS, Eten CB, Munteanu M, Loken MR, Van Dongen JJ, Bernstein ID, Appelbaum FR; Mylotarg Study Group. Antibody-targeted chemotherapy of older patients with acute myeloid leukemia in first relapse using Mylotarg (gemtuzumab ozogamicin). Leukemia. 2002 Sep;16(9):1627-36. doi: 10.1038/sj.leu.2402677. PMID 12200674
- [Background] Sievers EL, Larson RA, Stadtmauer EA, Estey E, Lowenberg B, Dombret H, Karanes C, Theobald M, Bennett JM, Sherman ML, Berger MS, Eten CB, Loken MR, van Dongen JJ, Bernstein ID, Appelbaum FR; Mylotarg Study Group. Efficacy and safety of gemtuzumab ozogamicin in patients with CD33-positive acute myeloid leukemia in first relapse. J Clin Oncol. 2001 Jul 1;19(13):3244-54. doi: 10.1200/JCO.2001.19.13.3244. PMID 11432892
- [Derived] Hibma J, Knight B. Population Pharmacokinetic Modeling of Gemtuzumab Ozogamicin in Adult Patients with Acute Myeloid Leukemia. Clin Pharmacokinet. 2019 Mar;58(3):335-347. doi: 10.1007/s40262-018-0699-5. PMID 30062662